CLINICAL TRIAL: NCT01829438
Title: Influence of a Distractive Auditory Stimulus on 6 Minute Walking Test in Healthy Children
Brief Title: Influence of Music on 6 Minutes Walking Distance in Healthy Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Principal Investigator, G.Reychler, Doctor in Physiotherapy, Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: 6MWT
Record Dates: First submitted 2013-04-09; First posted 2013-04-11 (Estimated); Last update posted 2013-04-11 (Estimated); Status verified 2013-04

CONDITIONS: Healthy Children
Keywords: exercise tolerance; 6MWT

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Without music (No Intervention): 6MWT without music
- With fast music (Experimental): 6MWT with a fast music
  Interventions: Behavioral: Listening to fast music
- With slow music (Experimental): 6MWT with a slow music
  Interventions: Behavioral: Listening to slow music
- With preferred music (Experimental): 6MWT with the preferred music of the child
  Interventions: Behavioral: Listening to preferred music

INTERVENTIONS:
Behavioral: Listening to fast music
  Other Names: Listening to fast music during the test
  Arms: With fast music
Behavioral: Listening to preferred music
  Other Names: Listening to preferred music during the 6MWT
  Arms: With preferred music
Behavioral: Listening to slow music
  Other Names: Listening to preferred music during the 6MWT
  Arms: With slow music

SUMMARY:
To evaluate the effect of different distractive auditory stimuli (fast, slow and preferred) on 6 Minute Walking Test (6MWT) and the measured parameters (dyspnea, heart rate, oxygen saturation) in healthy children.

ELIGIBILITY:
Inclusion Criteria:

* the participation to the physical education program after the annual medical investigation

Exclusion Criteria:

* a lung disease
* an overweight
* a motor disability based on parent's answers to a questionnaire

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 97 (Actual)
Dates: Start 2010-06; Primary Completion 2010-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Walked distance | After 6 minutes
  The distance walked by subjects during a 6 minutes walking test

SECONDARY OUTCOMES:
Dyspnea | At the end of the 6MWT
  Dyspnea is measured by a visual analogue scale

OTHER OUTCOMES:
cardio-respiratory parameters | at the begining and the end of the 6MWT
  Heart rate and oxygen saturation are measured before and after the test

CONTACTS AND LOCATIONS:
Overall Officials: Lux Amandine, Student, Principal Investigator — UCL
Locations (1):
- UCL, Brussels, Belgium